CLINICAL TRIAL: NCT04227262
Title: EFFICACY OF LOWER EXTREMITY MIRROR THERAPY ON BALANCE IN CHILDREN WITH HEMIPLEGIC CEREBRAL PALSY: A Randomized Controlled Trail
Brief Title: Efficacy of Lower Extremity Mirror Therapy on Balance in Children With Hemiplegic Cerebral Palsy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: South Valley University (Other)
Responsible Party: Principal Investigator, Mohammed E. Ali, Ph. D Candidate., Assistant Lecturer, South Valley University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/002575
Record Dates: First submitted 2020-01-04; First posted 2020-01-13 (Actual); Last update posted 2020-01-13 (Actual); Status verified 2020-01

CONDITIONS: HEMIPLEGIC CEREBRAL PALSY
Keywords: cerebral palsy; balance; mirror therapy
MeSH Terms: conditions — Cerebral Palsy | interventions — Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: The children were assigned randomly into two equal groups. Group (a) control group received traditional physical therapy program. And group (b) study group received the same traditional physical therapy program in addition to mirror therapy three times / weak for three successful months.
Who Masked: Outcomes Assessor
Masking Description: Blinding process to participants and care providers was impossible due to the nature of intervention therapy. Data were analyzed by an impartial statistician (outcomes assessor), referring to each arm with an encoded name: Group A (control group) and Group B (study group).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- the control group (No Intervention): Group (a) control group received traditional physical therapy program.
- the study group (Experimental): group (b) study group received the same traditional physical therapy program in addition to mirror therapy three times / weak for three successful months.
  Interventions: Other: MIRROR THERAPY

INTERVENTIONS:
Other: MIRROR THERAPY — The children were instructed to sitting on chair and a mirror is placed in midsagittal plane of the child, with the normal limb in front of mirror and the affected limb is blocked so the patient see only the reflected movement of the sound limb (non affected).
  Arms: the study group

SUMMARY:
The study will be conducted to assess the efficacy of mirror therapy on balance in children with hemiplegic cerebral palsy.

DETAILED DESCRIPTION:
Hemiplegic cerebral palsy in the most common type of cerebral palsy that has permanent motor disorders and associated with life-long disability. the aim of study to assess the efficacy of mirror therapy on balance in children with hemiplegic cerebral palsy. Seventy child with hemiplegic cerebral were enrolled in this study and were assessed for eligibility. Their aged ranged from eight to twelve years. The children were assigned randomly into two equal groups. Group (a) control group received traditional physical therapy program. And group (b) study group received the same traditional physical therapy program in addition to mirror therapy three times / weak for three successful months. Biodex balance system was used to assess balance pre and post treatment. All children were assisted before and after three months of intervention.

ELIGIBILITY:
Inclusion Criteria:

* Children's aged ranged from eight to twelve years.
* Children participated in this study will from both sexes.
* Their degree of spasticity will ranged from mild to moderate according to Modified Ashworth Scale.
* Children with stable medical and psychological status.
* Children able to follow the verbal commands or instructions.

Exclusion Criteria:

* children with visual or auditory problems.
* Children with history of epilepsy.
* Children with history of surgical interference in lower limbs less than one year.
* Medically unstable children especially with cardiovascular disorders.
* Mentally retarded children.
* un-cooperative children.

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 70 (Actual)
Dates: Start 2019-12-01 (Actual); Primary Completion 2020-03-01 (Estimated); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
Antro-posterior stability index | Antro-posterior stability index will be assessed at day 0.
  the ability of child to maintain his balance from forward to backward direction
Antro-posterior stability index | Antro-posterior stability index will be assessed at day 90.
  the ability of child to maintain his balance from forward to backward direction
Over All Stability Index | Over All Stability Index will be assessed at day 0.
  the ability of child to maintain his balance in all directions
Over All Stability Index | Over All Stability Index will be assessed at day 90.
  the ability of child to maintain his balance in all directions
Mediolateral Stability Index | Mediolateral Stability Index will be assessed at day 0.
  the ability of child to maintain his balance from side to side directions
Mediolateral Stability Index | Mediolateral Stability Index will be assessed at day 90.
  the ability of child to maintain his balance from side to side directions

CONTACTS AND LOCATIONS:
Overall Officials: Nehad A. Abo-zaid, PhD, Principal Investigator — South Valley University, Faculty of Physical Therapy; Mohammed E. Ali, PhD student, Principal Investigator — South Valley University, Faculty of Physical Therapy
Locations (1):
- South Valley University, Faculty of Physical Therapy, Qina, Qena Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gstottner M, Neher A, Scholtz A, Millonig M, Lembert S, Raschner C. Balance ability and muscle response of the preferred and nonpreferred leg in soccer players. Motor Control. 2009 Apr;13(2):218-31. doi: 10.1123/mcj.13.2.218. PMID 19454781
- [Background] Zeng W, Guo Y, Wu G, Liu X, Fang Q. Mirror therapy for motor function of the upper extremity in patients with stroke: A meta-analysis. J Rehabil Med. 2018 Jan 10;50(1):8-15. doi: 10.2340/16501977-2287. PMID 29077129
- [Background] Garry MI, Loftus A, Summers JJ. Mirror, mirror on the wall: viewing a mirror reflection of unilateral hand movements facilitates ipsilateral M1 excitability. Exp Brain Res. 2005 May;163(1):118-22. doi: 10.1007/s00221-005-2226-9. Epub 2005 Mar 8. PMID 15754176
- [Background] McInnes K, Friesen C, Boe S. Specific Brain Lesions Impair Explicit Motor Imagery Ability: A Systematic Review of the Evidence. Arch Phys Med Rehabil. 2016 Mar;97(3):478-489.e1. doi: 10.1016/j.apmr.2015.07.012. Epub 2015 Aug 5. PMID 26254950
- [Result] Kenis-Coskun O, Giray E, Eren B, Ozkok O, Karadag-Saygi E. Evaluation of postural stability in children with hemiplegic cerebral palsy. J Phys Ther Sci. 2016 May;28(5):1398-402. doi: 10.1589/jpts.28.1398. Epub 2016 May 31. PMID 27313338
- [Result] El-Shamy SM, Abd El Kafy EM. Effect of balance training on postural balance control and risk of fall in children with diplegic cerebral palsy. Disabil Rehabil. 2014;36(14):1176-83. doi: 10.3109/09638288.2013.833312. Epub 2013 Sep 13. PMID 24032716
- [Result] Altschuler EL, Hu J. Mirror therapy in a patient with a fractured wrist and no active wrist extension. Scand J Plast Reconstr Surg Hand Surg. 2008;42(2):110-1. doi: 10.1080/02844310701510355. PMID 18335358
- [Result] Funase K, Tabira T, Higashi T, Liang N, Kasai T. Increased corticospinal excitability during direct observation of self-movement and indirect observation with a mirror box. Neurosci Lett. 2007 May 29;419(2):108-12. doi: 10.1016/j.neulet.2007.04.025. Epub 2007 Apr 19. PMID 17481817
- [Result] Cattaneo L, Rizzolatti G. The mirror neuron system. Arch Neurol. 2009 May;66(5):557-60. doi: 10.1001/archneurol.2009.41. PMID 19433654
- [Result] Summers JJ, Kagerer FA, Garry MI, Hiraga CY, Loftus A, Cauraugh JH. Bilateral and unilateral movement training on upper limb function in chronic stroke patients: A TMS study. J Neurol Sci. 2007 Jan 15;252(1):76-82. doi: 10.1016/j.jns.2006.10.011. Epub 2006 Nov 28. PMID 17134723
- [Result] Sutbeyaz S, Yavuzer G, Sezer N, Koseoglu BF. Mirror therapy enhances lower-extremity motor recovery and motor functioning after stroke: a randomized controlled trial. Arch Phys Med Rehabil. 2007 May;88(5):555-9. doi: 10.1016/j.apmr.2007.02.034. PMID 17466722
- [Result] Saghaei M. Random allocation software for parallel group randomized trials. BMC Med Res Methodol. 2004 Nov 9;4:26. doi: 10.1186/1471-2288-4-26. PMID 15535880

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-01-03): https://cdn.clinicaltrials.gov/large-docs/62/NCT04227262/Prot_SAP_000.pdf